CLINICAL TRIAL: NCT00503893
Title: Genetics of Wilms' Tumor and/or the Associated Conditions of Aniridia, Hemihypertrophy, and Genitourinary Anomalies
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Other Study IDs: P80-099; P01CA034936-23 (NIH)
Record Dates: First submitted 2007-07-17; First posted 2007-07-19 (Estimated); Last update posted 2020-01-27 (Actual); Status verified 2020-01

CONDITIONS: Wilms' Tumor; Aniridia
Keywords: Wilms' Tumor; Genitourinary Anomalies; Beckwith-Wiedemann Hemihypertrophy; Aniridia; Questionnaire
MeSH Terms: conditions — Wilms Tumor; Aniridia; Urogenital Abnormalities | interventions — Surveys and Questionnaires; Blood Specimen Collection

STUDY DESIGN:
Observational Model: Family Based | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood sample(s) for genetic testing. Also, tissue samples, and/or bodily fluids (whether healthy or cancerous) left over from surgeries or procedures performed as part of standard care. The purpose of this clinical research study is to find out why some people develop cancers and tumors, why some families have more cancers than others, and whether certain genes or regions of DNA affect a person's risk of getting cancer.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Wilm's Tumor PO1: Familial and Sporadic Wilm's tumor, genitourinary anomalies, Beckwith-Wiedemann hemihypertrophy and/or aniridia.
  Interventions: Behavioral: Questionnaire; Other: Blood specimen

INTERVENTIONS:
Behavioral: Questionnaire — Questionnaire regarding medical history and family medical history that will take about 1 hour to complete.
  Other Names: Survey
Other: Blood specimen — Blood (about 10 teaspoons) will be drawn from a vein for genetic testing. The blood may be drawn more than one time.

SUMMARY:
The goal of this clinical research study is to collect information and blood samples to try to learn why some people develop cancers and tumors, why some families have more cancers than others, and whether certain genes or regions of DNA (the genetic material of cells) affect a person's risk of getting cancer.

This is an investigational study.

Up to 1500 patients and family members will take part in this study. All will be enrolled at MD Anderson.

DETAILED DESCRIPTION:
If you choose to take part in this study, blood (about 10 teaspoons) will be drawn for genetic testing. The blood may be drawn more than 1 time, depending on how much blood is drawn at the first visit, and if you are available for more blood draws. If this is the case, your doctor will discuss any extra blood draws with you.

For small children (less than 5 years old), about 2 teaspoons will be drawn. Children who are 5 years old or older will not have more than 3 teaspoons drawn.

You will complete a questionnaire about your medical history and family medical history. The questionnaire should take about 1 hour to complete. The study staff will also review your medical records.

You will be asked to allow the study staff to collect any of your tissue (whether healthy or cancerous) that is leftover from surgeries performed as part of your standard care. This may be from any past or future surgeries or any tissue being stored at MD Anderson or elsewhere. No new surgeries or biopsies will be performed for this study.

Before your information, tissue samples, and/or bodily fluids can be used for research, the people doing the research must get specific approval from the Institutional Review Board (IRB) of MD Anderson. The IRB is a committee made up of doctors, researchers, and members of the community. The IRB is responsible for protecting the participants involved in research studies and making sure all research is done in a safe and ethical manner. All research done at MD Anderson, including research involving your information, tissue samples, and/or bodily fluids, must first be approved by the IRB.

You may be contacted either by phone or mail 1 time a year, so that the study staff can update your medical history and information. If contacted by phone, this call should last about 30 minutes.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with familial and sporadic Wilm's tumor, genitourinary anomalies, Beckwith-Wiedemann hemihypertrophy and/or aniridia, and family members of patients.

Exclusion Criteria:

1. Patients who do not meet inclusion eligibility criteria are excluded.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Patients with familial and sporadic Wilm's tumor, genitourinary anomalies, Beckwith-Wiedemann hemihypertrophy and/or aniridia, and family members of patients.
Sampling Method: Non-Probability Sample
Enrollment: 295 (Actual)
Dates: Start 1980-12-01 (Actual); Primary Completion 2020-12 (Estimated); Study Completion 2020-12 (Estimated)

PRIMARY OUTCOMES:
Genetic Events Involved in Development of Wilms' tumor, Genitourinary Anomalies, Hemihypertrophy and Beckwith-Wiedemann, and/or Aniridia | 32 Years (Descriptive data collected using questionnaires)
  Characterize genetic events by a combined molecular biology/epidemiologic approach

CONTACTS AND LOCATIONS:
Overall Officials: Louise C. Strong, MD, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- University of Texas MD Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: University of Texas MD Anderson Cancer Center Website — http://www.mdanderson.org